CLINICAL TRIAL: NCT01385254
Title: Mother Sibling Interactions Following Very Low Birth Weight (VLBW) Infant Homecoming
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00019788; 1R03NR011196-01A1 (NIH)
Record Dates: First submitted 2011-01-20; First posted 2011-06-30 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Very Low Birthweight
Keywords: very low birthweight; premature; sibling adjustment; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- siblings and mothers of Very Low Birth Weight infants: 50 older siblings (closest in age) and mothers of very low birthweight (VLBW) infants, born at <33 weeks gestation and <1500 grams at birth
- siblings and mothers of healthy infants: 50 siblings (closest in age) and mothers of healthy, full-term infants (between 38-42 weeks gestation and lacking medical conditions that require a hospital stay past the mother's discharge date)

SUMMARY:
The proposed study will explore longitudinally the impact of a very low birthweight (VLBW) infant on mother-sibling interactions and sibling adjustment. The study will also include a comparison group of fullterm infants to determine which sibling adjustment problems are typical of having a new baby in the home and which are associated with the unique stress of having a VLBW infant. This study will be the initial step in identifying factors affecting the adjustment of siblings of VLBW infants.

DETAILED DESCRIPTION:
The proposed 2-year study will use a longitudinal, comparative, mixed method design to explore the impact of a Very Low Birth Weight (VLBW) (≤33 weeks gestational age) infant on mother-sibling interactions and sibling adjustment. A comparison group of full term infants (≥38 weeks gestational age) will be included to elucidate sibling adjustment problems that are typical to having a new baby in the home and sibling adjustment problems that are associated with the unique stress of having to care for a VLBW infant. Participants will be fifty mothers and siblings of VLBW infants and fifty mothers and siblings of full term infants. Data collection will take place within one week of infant discharge from the hospital (enrollment), and at 1 month and 6 months post infant discharge using self-report measures, qualitative interviews, and mother-sibling interaction observation. Variables of interest include mother's worry, anxiety, depression, and post-traumatic stress; mother-sibling interactions including uninvolvement, positive affect, negative affect, talk, looking and playing; internalizing and externalizing behaviors, sleep/somatic problems, and growth in siblings of VLBW and in siblings of the comparison group with full term infants. Mixed modeling and Ordinary Least Squares (OLS) regression modeling will be conducted to identify factors that make siblings vulnerable to psychological and emotional adjustment problems in response to having a VLBW infant in the home. There are no anticipated risks for the infant participants of the study aside from the small risk of violating confidentiality of infant participants and their mothers. No risks for siblings are anticipated aside from the small risk of violating confidentiality.

ELIGIBILITY:
Inclusion Criteria for siblings:

* Siblings of very low birth weight or healthy, full-term infants
* age 4 years old or younger
* siblings and infants must live with the mother

Inclusion Criteria for mothers:

* no previous or current diagnosis of major psychological disorder (including bipolar disorder, psychosis, or active substance abuse)
* age 18 years or older
* English speaking,
* living within 1 hour's travel distance from Duke University, for feasibility.
* Mothers at-risk for preterm birth who meet all other eligibility criteria

Exclusion Criteria:

Mother/sibling pairs of infants who:

* have congenital neurological problems (congenital hydrocephalus or microcephaly),
* are symptomatic from substance exposure,
* are hospitalized longer than 1 month after term, or
* are technology dependent.

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mothers who give birth at Duke University Medical Center, Durham Regional Hospital, or Wake Medical Center, and their siblings.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Differences in level of maternal worry in mothers of very low birthweight (VLBW) infants compared to mothers of full-term infants | baseline, one month, six months
  Explore how the trajectories of maternal worry about the infant and sibling, anxiety, depression, post traumatic stress, concerns for and expectations of the sibling, and perceptions of sibling growth over the 6-month post discharge period differ between mothers of VLBW infants and mothers of fullterms.
Differences in mother-sibling interaction between two groups | one month and six months
  Explore differences in mother-sibling interactions, including involvement, positive/negative affect, talking, looking and playing, at 1 and 6 months after infant discharge between the two groups of siblings and mothers, using a coding schema to score videotaped interactions.
Differences in internalizing and externalizing behaviors between two groups | one month and six months
  Explore differences in internalizing and externalizing behaviors, vulnerability, and sleep/somatic problems at 6-months post-infant discharge between siblings of VLBW infants and siblings of fullterms, using a coding schema to score videotaped interactions.

SECONDARY OUTCOMES:
Effects of maternal worry, anxiety, depression and Post-Traumatic Stress Disorder (PTSD) on two groups | one month and six months
  Examine the effects of maternal worry, anxiety, depression, and post traumatic stress on group differences in mother-sibling interactions at 1 and 6 months after infant discharge.
Change in mother-sibling interactions between groups | one month and six months
  Examine the effects of changes in mother-sibling interactions from 1 to 6 months after infant discharge on group differences in siblings' internalizing and externalizing behaviors, vulnerability, and sleep/somatic problems.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Thompson, PhD, Principal Investigator — Duke University School of Nursing
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Wake Medical Center, Raleigh, North Carolina